CLINICAL TRIAL: NCT01253408
Title: Study of the Effect of Cannabinoid Agonist on Gastrointestinal and Colonic Motor and Sensory Functions in Patients With Irritable Bowel Syndrome
Brief Title: Effect of Cannabinoid Agonist on Gastrointestinal and Colonic Motor Functions in Patients With Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Dr. Michael Camilleri, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 08-008314 Part A; R01DK079866 (NIH); UL1RR024150 (NIH)
Record Dates: First submitted 2010-11-18; First posted 2010-12-03 (Estimated); Results first posted 2013-05-07 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: anandamide; cannabinoid; fatty acid amide hydrolase; gastric; motility; small bowel
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dronabinol 2.5 mg bid (Experimental): Dronabinol 2.5 mg will be taken orally with water twice per day for two days.
  Interventions: Drug: Dronabinol
- Dronabinol 5 mg bid (Experimental): Dronabinol 5 mg will be taken orally with water twice per day for two days.
  Interventions: Drug: Dronabinol
- Placebo (Placebo Comparator): Placebo will be taken orally with water twice per day for two days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol — Dronabinol is a synthetic delta-9-tetrahydrocannabinol, a nonselective cannabinoid agonist. Subjects will receive either 2.5 mg bid, or 5 mg bid, taken orally with water for 2 days.
  Other Names: Marinol
  Arms: Dronabinol 2.5 mg bid; Dronabinol 5 mg bid
Drug: Placebo — Placebo will match study drug; taken orally with water twice per day for two days.
  Arms: Placebo

SUMMARY:
Irritable bowel syndrome (IBS) affects about 15% of the U.S. population. There are still no effective and safe medications approved for the treatment of abdominal pain associated with bowel symptoms in IBS. This study will investigate the effects of an approved medication, Dronabinol, on the movement of food through the stomach and colon in subjects with a history of diarrhea-predominant Irritable Bowel Syndrome (D-IBS).

Dronabinol is a synthetic medication (a medication made in a laboratory) related to the active ingredient of "cannabinoid or marijuana". Dronabinol is approved by the Food and Drug Administration (FDA) for preventing nausea and vomiting in patients with cancers undergoing chemotherapy. It is also used in AIDS patients with excessive weight loss for improvement in appetite and weight gain.

The hypothesis in this study is that dronabinol will slow down the movement of food through the colon, and that this effect is regulated by the genes controlling the body messengers (receptors) that respond to medicinal marijuana or synthetic medicines that work on the same messengers that are present in the gastrointestinal tract and pain nerves.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) affects about 15% of the U.S. population. Despite increasing understanding of the pathophysiology of IBS, there are unmet clinical needs and no effective medication approved for the treatment of abdominal pain associated with IBS. Cannabinoid receptors (CBR) are on cholinergic neurons in the brain stem, stomach and colon. A cannabinoid receptor type 1 (CB1) antagonist, rimonabant, is effective in induction of weight loss; however, the mechanism of this benefit is unclear. Human studies from this lab show that a CBR agonist, dronabinol, inhibits gastric and colonic motility, which may alter appetite or satiation in obesity, and may have potential in the treatment of IBS. The overall focus of the study is on the mechanisms involved in the modulation of gastric and colonic motor and sensory functions by cannabinoid receptors (CBR) in health and in IBS. CB1 receptors are also involved in nociception and in mediating inflammation which are increasingly recognized as being potential pathophysiological mechanisms in IBS. The aims of the study are to compare the effects of two doses of the cannabinoid agonist, dronabinol (5 and 10 mg/day) and placebo on gastrointestinal and colonic motor and sensory functions in IBS. Also, to determine whether variations in the fatty acid amide hydrolase (FAAH) gene and the monoacylglycerol lipase (MGLL) gene (for the rate limiting enzyme, monoacylglycerol lipase, for another endocannabinoid, 2-arachidonyl glycerol) influence the pharmacological effect of cannabinoid modulation on gastrointestinal motor and sensory functions.

All participants underwent the following procedures:

1. Documentation of eligibility, screening questionnaires, and physical examination within the month prior to the study. The physical exam included standard rectal and pelvic floor examinations to exclude rectal evacuation disorder. This was necessary to ensure the diarrhea ws not secondary to "retention of stool with overflow."
2. Baseline colonic transit measurement (Geometric Center 24-h and 48-h), off treatment.
3. Treatment days corresponded to the scintigraphic transit testing days (days 1 and 2) with participants receiving the medication to which they were randomized. Scintigraphic measurements of gastric, small bowel, and colonic transit were conducted, using a previously validated method on days 1 and 2, and were completed with a fasting 48-h scan on day 3 when no medication was administered.

   On days 1 and 2, the morning dose of medication was ingested in the research laboratory, with the participant fasting. On day 1, the morning dose of medication was administered together with the delayed release capsule containing an isotope labeled activated charcoal used to measure colonic transit. On day 2, the morning dose of medication was given after the 24-h scan. The evening doses on days 1 and 2 were ingested by participants at bed time in their homes.
4. With appropriate consent, a venous blood sample was to be obtained from all participants for DNA extraction and pharmacogenomic studies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Positive for IBS symptoms by Rome III criteria
* No prior abdominal surgery (except appendectomy or cholecystectomy)
* Baseline Geometric Center at 24 hours is greater/equal to 2.0
* Baseline Geometric Center at 48 hours is greater/equal to 3.9

Exclusion Criteria:

* Patients with significant depression (score of greater than 10 on Hospital and Anxiety Inventory)
* Patients with anxiety (score of greater than 10 on Hospital and Anxiety Inventory) will not be allowed to participate. However, patients on stable doses of selective serotonin re-uptake inhibitors (SSRIs) or low dose of tricyclic antidepressants will be eligible.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Wong BS, Camilleri M, Busciglio I, Carlson P, Szarka LA, Burton D, Zinsmeister AR. Pharmacogenetic trial of a cannabinoid agonist shows reduced fasting colonic motility in patients with nonconstipated irritable bowel syndrome. Gastroenterology. 2011 Nov;141(5):1638-47.e1-7. doi: 10.1053/j.gastro.2011.07.036. Epub 2011 Jul 29. PMID 21803011
- [Result] Wong BS, Camilleri M, Eckert D, Carlson P, Ryks M, Burton D, Zinsmeister AR. Randomized pharmacodynamic and pharmacogenetic trial of dronabinol effects on colon transit in irritable bowel syndrome-diarrhea. Neurogastroenterol Motil. 2012 Apr;24(4):358-e169. doi: 10.1111/j.1365-2982.2011.01874.x. Epub 2012 Jan 30. PMID 22288893

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited from a database of patients with irritable bowel syndrome (IBS) who reside within 150 miles of Rochester, Minnesota from October 2008 through April 2011.
Period: Overall Study
Arm/Group | Dronabinol 2.5 mg Bid | Dronabinol 5 mg Bid | Placebo
Started | 10 | 13 | 13
Completed | 10 | 12 | 13
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dronabinol 2.5 mg Bid | Dronabinol 5 mg Bid | Placebo | Total
Number analyzed (Participants) | 10 | 13 | 13 | 36
Age Continuous [Mean (Standard Deviation); unit: years] | 47.68 (25.08) | 42.28 (16.36) | 36.7 (11.02) | 41.77 (17.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 13 | 34
  Male | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 13 | 13 | 36
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.7 (1.5) | 31.6 (3.9) | 30.8 (1.8) | 30.50 (9.46)

OUTCOME MEASURES:

1. Secondary Outcome: Colonic Transit Geometric Center
Description: The scintigraphic method is used to measure colonic transit. An isotope is adsorbed on activated charcoal particles and delivered to the colon in a delayed release capsule. Anterior and posterior gamma images are taken hourly. The geometric center (GC) is the weighted average of counts in the different colonic regions. The scale ranges from 1 to 5; a high GC implies faster colonic transit, a GC of 1 implies all isotope is in the ascending colon, and a GC of 5 implies all isotope is in the stool.
Time Frame: 28, 32, and 48 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dronabinol 2.5 mg Bid | Dronabinol 5 mg Bid | Placebo
Number analyzed (Participants) | 10 | 13 | 13
units on a scale
  28 hours | 3.39 (1.28) | 3.60 (1.04) | 3.24 (1.18)
  32 hours | 3.78 (1.11) | 4.05 (0.90) | 3.54 (1.17)
  48 hours | 4.21 (0.94) | 4.60 (0.65) | 4.02 (0.99)

2. Secondary Outcome: Gastric Emptying Half-Time (t1/2)
Description: The time for half of the ingested solids or liquids to leave the stomach.
Time Frame: Approximately 2 hours after radiolabel meal is ingested
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Dronabinol 2.5 mg Bid | Dronabinol 5 mg Bid | Placebo
Number analyzed (Participants) | 10 | 13 | 13
minutes | 137.3 (33.53) | 130.7 (42.13) | 138.2 (45.18)

3. Secondary Outcome: Colonic Filling at 6 Hours
Description: Percent of the radio-labeled meal that reached the colon at 6 hours, indirectly reflecting small bowel transit time.
Time Frame: 6 hours after radiolabeled meal was ingested
Measure: Mean (Standard Deviation); unit: percentage of meal
Arm/Group | Dronabinol 2.5 mg Bid | Dronabinol 5 mg Bid | Placebo
Number analyzed (Participants) | 10 | 13 | 13
percentage of meal | 48.60 (33.76) | 51.62 (29.89) | 57.46 (24.77)

4. Secondary Outcome: Ascending Colon Emptying T 1/2
Description: Ascending colon emptying t1/2 will be estimated by power exponential analysis of the proportionate emptying over time of counts from the colon. The primary data for this analysis will be the proportion of decay and depth-corrected counts in the ascending colon on the hourly scans on the first day of transit measurement and the 48 hour data.
Time Frame: 48 hours after radiolabeled meal was ingested
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dronabinol 2.5 mg Bid | Dronabinol 5 mg Bid | Placebo
Number analyzed (Participants) | 10 | 13 | 13
hours | 9.50 (4.62) | 9.90 (5.44) | 14.53 (8.36)

5. Secondary Outcome: Gastric Emptying at 2 and 4 Hours
Description: Proportion of stomach contents emptied at a 2 and 4 hours.
Time Frame: 2, 4 hours
Measure: Mean (Standard Deviation); unit: proportion of stomach contents
Arm/Group | Dronabinol 2.5 mg Bid | Dronabinol 5 mg Bid | Placebo
Number analyzed (Participants) | 10 | 13 | 13
proportion of stomach contents
  2 hours | 0.38 (0.15) | 0.49 (0.17) | 0.45 (0.14)
  4 hours | 0.90 (0.09) | 0.90 (0.13) | 0.88 (0.16)

6. Primary Outcome: Colonic Transit Geometric Center at 24 Hours
Description: as for outcome 1
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dronabinol 2.5 mg Bid | Dronabinol 5 mg Bid | Placebo
Number analyzed (Participants) | 10 | 13 | 13
units on a scale | 3.12 (1.29) | 3.05 (1.02) | 2.77 (1.23)

ADVERSE EVENTS:
Arm/Group | Dronabinol 2.5 mg Bid | Dronabinol 5 mg Bid | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 7/10 | 9/13 | 7/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dronabinol 2.5 mg Bid (N=10) | Dronabinol 5 mg Bid (N=13) | Placebo (N=13)
Hot flushing (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Headache (General disorders) | 3 (3) | 2 (2) | 2 (2)
Dizziness/lightheadedness (General disorders) | 2 (2) | 4 (4) | 1 (1)
Drowsiness/tiredness (General disorders) | 4 (4) | 5 (5) | 4 (4)
"Loopy," foggy thinking (General disorders) | 1 (1) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
This study included assessment of only four doses of dronabinol over 2 days.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No